CLINICAL TRIAL: NCT00183976
Title: A Pilot Phase II Study of Pegylated Liposomal Doxorubicin (Doxil) With Rituximab in Relapsed AIDS-Related Non-Hodgkin's Lymphomas
Brief Title: Pegylated Liposomal Doxorubicin (Doxil) With Rituximab in Relapsed AIDS-Related Non-Hodgkin's Lymphomas
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient Accrual
Sponsor: University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17NHL-03-2
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2006-05

CONDITIONS: Non-Hodgkin's Lymphoma; Burkitt Lymphoma; Primary Effusion Lymphomas
Keywords: Diffuse mixed NHL; Diffuse or follicular large B-cell NHL; Immunoblastic NHL; Burkitt or Burkitt-like lymphomas
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Burkitt Lymphoma; Lymphoma, Primary Effusion | interventions — liposomal doxorubicin; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Pegylated Liposomal Doxorubicin (Doxil) and Rituximab

SUMMARY:
This study is for patients who have been treated before and either the treatment did not work or the lymphoma has come back.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented B-cell non-Hodgkin's lymphoma [NHL] (diffuse mixed, diffuse or follicular large B-cell, immunoblastic), Burkitt or Burkitt-like lymphomas, and primary effusion lymphomas.
* Seropositive for HIV by any approved test (prior documentation of HIV seropositivity is acceptable).
* Failed or relapsed after at least 1 prior chemotherapy treatment (chemotx) regimen but could have had no more than 2 prior chemotx regimens with only one of them being an anthracycline-containing regimen. Prior treatment (tx) with rituximab allowed.
* All stages of disease
* Measurable or evaluable tumor
* Greater than or equal to 18 years of age
* Karnofsky performance status greater than 50%
* Absolute granulocyte count (AGC) greater than 1.0; platelets greater than 75,000; hemoglobin (Hgb) greater than 8.0 (unless these parameters are abnormal secondary to lymphomatous involvement of marrow, or due to HIV-related thrombocytopenia).
* Bilirubin less than 2.0 (unless elevated secondary to lymphomatous involvement of liver or biliary system or due to other HIV-related medications such as Crixivan).
* Creatinine less than 2.5 or creatinine clearance greater than 60 ml/min
* Multigated acquisition (MUGA) scan or 2D echocardiogram indicating left ventricular ejection fraction (LVEF) greater than or equal to 50% within 42 days prior to first dose of study drug.
* Patients with central nervous system (CNS) involvement are eligible provided that systemic lymphomatous disease is also present.
* Concurrent therapy for HIV with any licensed agent or an agent available on an expanded access program will be required.
* Signed informed consent including Health Insurance Portability and Accountability Act of 1996 (HIPAA) authorization.

Exclusion Criteria:

* Acute intercurrent infection that may interfere with planned protocol. Patients with mycobacterium avium are not excluded. Chronic therapy with potentially myelosuppressive agents is allowed provided that entry hematologic criteria are met.
* Second active tumor. Patients with non-melanomatous skin cancer, in-situ cervical cancer, or Kaposi's sarcoma, not requiring systemic chemotherapy may be entered on study.
* Primary CNS lymphoma.
* Documented history of congestive heart failure (CHF), hemodynamically unstable arrhythmia, myocardial infarction (MI) in the preceding 6 months, or evidence on electrocardiogram (EKG) of untreated cardiac ischemia.
* Prior exposure to a liposomal anthracycline (liposomal doxorubicin or daunorubicin) for the treatment of lymphoma. Prior exposure to conventional doxorubicin allowed.
* Prior radiation therapy within 4 weeks, unless for emergency conditions secondary to lymphoma (i.e., CNS tumor, cord compression)
* Prior systemic chemotherapy or biologic therapy within 3 weeks
* History of hypersensitivity reaction to anthracyclines or granulocyte colony-stimulating factor (G-CSF)
* History of hypersensitivity reactions attributed to a conventional formulation of doxorubicin hydrochloride (HCl)
* Investigational agent(s) within 4 weeks of start of study therapy.
* History of cardiac disease with New York Heart Association (NYHA) greater than or equal to Class II, or clinical evidence of CHF
* Pregnant or nursing mothers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2005-04; Primary Completion 2005-09 (Actual); Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anil Tulpule, MD, Principal Investigator — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California, United States